CLINICAL TRIAL: NCT06818591
Title: Preventive Effect of Helicobacter Pylori Eradication on Osteoporosis in Females: Prospective Observational Cohort Study for Up to 20 Years
Brief Title: Preventive Effect of H.Pylori Eradication on Osteoporosis
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2401-878-002
Record Dates: First submitted 2025-02-03; First posted 2025-02-10 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: HELICOBACTER PYLORI INFECTIONS; Osteoporosis
Keywords: Helicobacter pylori eradication; osteoporosis; Sex difference; Age
MeSH Terms: conditions — Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Eradicated group: Helicobacter pylori eradication was successfully achieved.
  Interventions: Diagnostic Test: DEXA(Dual-Energy X-ray Absorptiometry)
- Non-eradicated group: Helicobacter pylori eradication was not successfully achieved.
  Interventions: Diagnostic Test: DEXA(Dual-Energy X-ray Absorptiometry)

INTERVENTIONS:
Diagnostic Test: DEXA(Dual-Energy X-ray Absorptiometry) — Followed for up to 20 years

SUMMARY:
In this study, the investigators observed the long-term incidence rate of osteoporosis in patients who received Helicobacter pylori eradication and examined differences by age and sex.

DETAILED DESCRIPTION:
In this study, the investigators observed the long-term incidence rate of osteoporosis in patients who received Helicobacter pylori eradication and examined differences by age and sex. In addition, the investigators will analyze the correlation between the incidence of osteoporosis by comparing confounding factors such as body mass index, steroid use, and proton pump inhibitor use as well as the eradication status of H. pylori.

ELIGIBILITY:
Inclusion Criteria:

ㆍPatients tested Helicobacter pylori status

Exclusion Criteria:

ㆍPatients aged < 20 years ㆍPatients with unknown Helicobacter pylori bone density status ㆍPatients with with a history of gastric cancer ㆍPatients with prior Helicobacter pylori eradication therapy ㆍPatients with a history of osteoporosis

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients tested Helicobacter pylori status in Seoul National University Bundang Hospital, from 2003 to 2023
Sampling Method: Non-Probability Sample
Enrollment: 846 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2023-02 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
the incidence of new-onset osteoporosis | The patients were prospectively monitored until they either developed osteoporosis or reached the study endpoint in February 2023, whichever occurred first.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim Y, Choi Y, Kim N, Jeon EB, Kong SH, Lee JH, Lee HK, Jun YK, Yoon H, Shin CM, Park YS, Lee DH, Ahn S. Preventive Effect of Helicobacter pylori Eradication on Osteoporosis in Females: A 20-Year Prospective Observational Cohort Study. Gut Liver. 2025 Aug 18. doi: 10.5009/gnl250164. Online ahead of print. PMID 40820207